CLINICAL TRIAL: NCT06445738
Title: A Two-arm, Non-randomised, Prospective, Multicentre Study Using Magnetic Resonance Imaging (MRI) Findings and Pathology Features to Select Patients With Early Breast Cancer for Omission of Post-operative Radiotherapy
Brief Title: Post-operative Radiotherapy Omission in Selected Patients With Early Breast Cancer Trial International VErsion (PROSPECTIVE)
Acronym: PROSPECTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Breast Cancer Trials, Australia and New Zealand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BCT 2401
Record Dates: First submitted 2024-05-24; First posted 2024-06-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Cancer Female
Keywords: Omission of radiotherapy; Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A two-arm, non-randomised, prospective, multicentre study using MRI findings and pathology features to select patients with early breast cancer for omission of post-operative radiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy Omission (Experimental): Participants with nil, minimal or mild parenchymal enhancement on pre-operative MRI whose pathology meets inclusion/exclusion requirements for omission of post-operative radiotherapy will be allocated to Arm A, unless the participant prefers to receive Standard Treatment (Arm B) or following clinical team recommendation.
  Arm A participants will be divided into 2 groups:
  * Arm A1: Grade 1 or 2/HER2 negative ("low risk")
  * Arm A2: Grade 3 and/or HER2 positive ("high risk")
  Interventions: Radiation: Arm A: Radiotherapy Omission
- Standard Treatment (Active Comparator): Participants who are found to be ineligible for RT omission on study; includes management of MRI-detected lesions.
  Participants with any of:
  * Moderate or marked parenchymal enhancement on pre-operative MRI
  * A malignant occult lesion identified on MRI; or
  * Pathology that does not meet inclusion/exclusion criteria will receive standard multidisciplinary team recommendations to guide treatment. Participants may also be included in Arm B due to their own preference or following clinical team recommendation.
  Interventions: Other: Arm B: Standard Treatment

INTERVENTIONS:
Radiation: Arm A: Radiotherapy Omission — Omission of radiotherapy based on pre-surgical MRI and pathology findings at surgery.
  Other Names: A1: Grade 1 or 2/HER2 negative; A2: Grade 3 and/or HER2 positive
  Arms: Radiotherapy Omission
Other: Arm B: Standard Treatment — Ineligible for RT omission on study; includes management of MRI-detected lesions.
  Arms: Standard Treatment

SUMMARY:
The PROSPECTIVE trial aims to find out if using the results of Magnetic Resonance Imaging (MRI) for early breast cancer can select people to not have radiotherapy and still have a low chance of the cancer coming back after surgery.

The main question it aims to answer is:

* Will cancer come back in the same breast as the original cancer in patients who have surgery for their breast cancer, but who don't have radiotherapy afterwards because the results of an MRI before surgery showed favourable characteristics for not having radiotherapy.

DETAILED DESCRIPTION:
Breast cancer is the most common serious malignancy in women and most patients are suitable for therapy involving surgery and adjuvant radiotherapy (RT). For most patients, there is a lack of evidence that breast conserving surgery without adjuvant RT is safe and therefore patients bear the costs, inconvenience and morbidity of RT. Prior attempts to identify large subsets of patients for whom RT can be safely omitted based on clinicopathological features of the index cancer have had limited success, and so RT is currently omitted only in some women over 65 or 70 with small low risk cancers. Identification of a much larger subset of patients in whom adjuvant RT could be safely omitted would be hugely significant, not only to the patients, but to the entire health system.

The ANZ 1002 PROSPECT study was a two-arm phase II study that used breast MRI findings and pathological features to identify a group of patients with low risk early breast cancer in whom RT may be safely omitted. The findings at the primary strongly support the hypothesis and suggest that the combination of preoperative MRI and pathological features can identify a substantial group of early breast cancer patients in whom adjuvant RT can be safely omitted.

A Health Economic analysis of PROSPECT found that the avoided costs of RT and its potential side effects is likely to substantially outweigh the extra cost of MRI scans and associated investigations. Parallel cross-sectional studies assessing Fear of Cancer Recurrence (FCR) and Health Related Quality of Life (HRQoL) in patients taking part in PROSPECT who either did or did not receive RT and a control group found a substantially lower FCR in PROSPECT patients who omitted RT as well as improved HRQoL.

The majority of screened and eligible patients (427/443 and 193/201, respectively) for PROSPECT were recruited from two Australian sites. Before the PROSPECT approach can be widely adopted, the findings need to be replicated in a multicentre, international study. In addition, patient reported outcomes and health economic assessments need to be performed prospectively and longitudinally.

PROSPECTIVE is the follow-up to PROSPECT which will address these issues, and also include translational research aspects to further study the natural history and outcomes of this group of lower risk early breast cancers.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study at Registration, participants must fulfil all of the following criteria:

1. Has provided written, informed consent to participate in the study.
2. Female participants ≥ 50 years old with histologically* confirmed ER-positive and/or HER2-positive invasive breast cancer.
3. Has a life expectancy of at least 10 years and suitable for prolonged follow up for 10 years.
4. Breast imaging indicating unifocal, unilateral breast cancer must have been performed before pre-registration.
5. Willing/able to have surgery within 8 weeks of registration or pre-operative MRI, whichever occurs later.
6. Have ECOG performance status 0-2.

   * Oestrogen receptor and progesterone receptor status of invasive cancer will be assessed by immunohistochemistry on the diagnostic core biopsy specimen. The IHC results will be reported as percentage of nuclei stained and a score of intensity from negative, weak, intermediate or high staining

HER2 neu status will be assessed by immunohistochemistry and will be scored as follows46:

* 0 or 1+ (HER2 negative): No staining or membrane staining that is incomplete and is faint/barely perceptible and in ≤ 10% of tumour cells (0); or incomplete membrane staining that is faint/barely perceptible and in > 10% of tumour cells (1+).
* 2+ (equivocal): weak to moderate complete membrane staining observed in > 10% of tumour cells. Must order reflex test (same specimen using ISH) or order a new test (new specimen if available using HIS or ISH).
* 3+ (HER2 positive): Circumferential membrane staining that is complete, intense and in > 10% of tumour cells.

Exclusion Criteria:

Any one of the following at Registration is regarded as a criterion for exclusion from the study:

1. Triple negative breast cancer (ER-negative and PR-negative and HER2-negative) where ER and PR positivity is defined as ≥ 10% staining on IHC.
2. Previous invasive breast cancer and/or DCIS in either breast.
3. Prior RT to the breast or chest.
4. Participants who plan to have a mastectomy for the index cancer.
5. Lymphovascular invasion (LVI) reported on diagnostic core biopsy.
6. Multifocal/multicentric breast cancer on breast imaging before registration.
7. Distant metastasis at diagnosis.
8. Bilateral breast cancer
9. Known breast cancer predisposition gene mutation carriers (BRCA1, BRCA2, PALB2, CHEK2, ATM, CDK1, p53, BARD1, RAD51C, RAD51D, CDH1, STK11, PTEN).
10. Contraindication to breast MRI scanning.
11. Concurrent illness/conditions which limits life expectancy to 10 years or less.
12. Has moderate or marked BPE in the breast containing the index cancer (where MRI is done before registration).
13. Inability to give informed consent.

Allocation: Arm A - Radiotherapy Omission

In addition to the above criteria, for inclusion in the omission of radiation therapy arm of the study after surgery, participants must fulfil all the following criteria. Participants not fulfilling any one of the following criterial will be allocated to Arm B:

1. Has nil/minimal or mild BPE in the breast containing the index lesion on pre-operative breast MRI.
2. BCS with unifocal**, invasive primary tumour (including any surrounding DCIS) ≤ 20 mm.

   The overall tumour size (including additional foci of DCIS) must remain ≤ 20 mm. The tumour size is defined as the longest distance between the outer most edges of all foci, the space between the two or more foci is included in the overall size: Size = ('Focus A + Focus B + 'the distance between A and B').
3. Radial resection margins must be ≥ 2 mm clear of any invasive cancer and ≥ 2 mm clear of any DCIS. Superficial or deep margins of < 2 mm for invasive cancer and DCIS are allowed if there is no tumour on ink and all breast tissue from the subcutaneous tissue or pectoralis fascia respectively was removed and radial margins are ≥ 2 mm for invasive cancer and DCIS.
4. pN0 (pN0 i+ is eligible for inclusion) by sentinel node biopsy and/or axillary dissection.
5. Absence of LVI and extensive intraductal component (EIC) on final pathology.
6. The extent of invasive cancer is at least 50% of the total tumour size (invasive cancer + DCIS).
7. Have no additional BIRADS 3+ lesions not shown to be benign on pre-operative or surgical biopsy.
8. Participants with Grade 3 cancer and/or HER2-positive cancer must agree to comply with systemic treatment recommendations.
9. Participants must be allocated to a treatment arm within 8 weeks after final breast surgery.

   * Where histopathology is unable to identify a 'bridge' of tumour tissue joining two or more apparent invasive cancer foci the following will be used to confirm unifocal disease:

     * All foci must be of the same histological subtype
     * All foci must have the same hormone (ER and PR) and HER2 status.

Allocation: Arm B - Standard Treatment (ineligible for RT omission on study; includes management of MRI-detected lesions)

In addition to the above Inclusion Criteria, participants who fulfil one any of the following criteria will receive standard treatment:

1. Has moderate or marked BPE in the breast containing the index lesion on pre-operative breast MRI.
2. Has a biopsy-proven mOL identified on breast MRI.
3. Suspicious lesion identified on CEM but not on MRI and confirmed on investigation to be a DCIS or invasive breast cancer.
4. Surgical pathology does not meet the inclusion criteria. 2mm radial margins are required, as guidelines suggesting "no tumour on ink" relate to those receiving adjuvant RT.
5. Clinical team meeting determination that RT be recommended.
6. Participant chooses to have RT despite being eligible for RT omission.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2039-06 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral Invasive Recurrence Rate (IIRR) in low-risk patients omitting RT at a median of 5 years follow up | Median of 5 years follow up (when 300th low risk patient in Arm A reaches 5 years follow up)
  To determine the ipsilateral invasive recurrence rate (IIRR) in lower risk patients with unequivocally unifocal breast cancer and on breast MRI and favourable clinico-pathological features.

SECONDARY OUTCOMES:
Ipsilateral Invasive Recurrence Rate (IIRR) in all participants omitting RT at a median of 10 years follow up after surgery. | Median of 10 years follow up after surgery.
  To determine the ipsilateral invasive recurrence rate (IIRR) in patients allocated to omit radiotherapy (Arm A1).
IIRR in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B. | Median of 5 years and 10 years follow up after surgery.
  To determine the ipsilateral invasive recurrence rate (IIRR) in participants in Arm A2, Arm A, Arm B, and Arms A+B.
Ipsilateral DCIS recurrence rate in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B. | Median of 5 and 10 years follow up after surgery.
  To determine the ipsilateral DCIS rate in the breast in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B.
The combined ipsilateral DCIS and invasive recurrence rate (IRR) in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B. | Median of 5 and 10 years follow up after surgery.
  To determine the combined ipsilateral DCIS and invasive recurrence rate (IRR) in the breast in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B.
Regional recurrence rate in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B. | Median of 5 and 10 years follow up after surgery.
  To determine the regional recurrence rate in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B.
Distant recurrence rate in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B.. | Median of 5 and 10 years follow up after surgery.
  To determine the distant recurrence rate in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B.
Contralateral DCIS and invasive breast cancer rate in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B | Median of 5 and 10 years follow up after surgery.
  To determine the contralateral DCIS and invasive breast cancer rate in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B.
Breast cancer specific survival (BCSS) in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B | Median of 5 and 10 years follow up after surgery.
  BCCS rate defined as the percentage of people who have not died from breast cancer.
Overall Survival (OS) in participants in Arm A1, Arm A2, Arm A, Arm B, and Arms A+B. | Median of 5 and 10 years follow up after surgery.
  OS rate defined as the percentage of people alive.
PRO: Fear of Cancer Recurrence | Median 24 months post-surgery
  To determine the difference in Fear of cancer recurrence (FCR) between Arm A and Arm B measured by the Fear of Cancer Recurrence Inventory Short Form (FCRI-SF). A higher score indicates a greater fear of recurrence.
PRO: Levels of FCR and perception of risk of recurrence in Arm A over time. | At median of 24 months post-surgery
  To determine the difference in levels of FCR and perception of risk of recurrence in Arm A measured by the Fear of Cancer Recurrence Inventory - Short Form and 2 items adapted from Abbott et al. A higher score indicates greater fear of recurrence and greater risk perception.
PRO: Difference in FCR and perception of risk of recurrence between Arm A and Arm B. | From allocation to 3-, 6-, 12-, 24- and 60 months median follow-up post-surgery.
  To determine the difference over time in FCR and perception of risk of recurrence between Arm A and Arm B over time as measured by the FCRI-SF and 2 items adapted from Abbott et al. A higher score indicates greater fear of recurrence and greater risk perception.
PRO: Perception of risk of recurrence in Arm A and between Arm A and Arm B. | From allocation to 3-, 6-, 12-, 24- and 60 months median follow up post-surgery
  To determine the difference in perceptions of risk of recurrence in the breast and elsewhere in the body measured by 2 items adapted from Abbott et al. A higher score indicates greater risk perception.
PRO: Health Related Quality of Life (HRQoL) (functional and aesthetic outcomes, fatigue, body image, financial toxicity) between Arm A and Arm B. | At a median of 24 months post-surgery.
  To determine the difference in breast-specific symptoms, cosmetic status, arm- and shoulder functional status measured by the Breast Cancer Treatment Outcomes Scale (BCTOS); and fatigue, body image, financial toxicity measured by the EORTC IL353. A higher score indicates greater morbidity, greater fatigue; greater financial toxicity; poorer body image.
PRO: Health Related Quality of Life (HRQoL) (functional and aesthetic outcomes, fatigue, body image, financial toxicity) in Arm A | From allocation to 3-, 6-, 12-, 24- and 60 months median follow up post-surgery
  To determine the HRQoL (functional and aesthetic outcomes, fatigue, body image, financial toxicity), in Arm A measured by the BCTOS (breast-specific symptoms, cosmetic status, arm- and shoulder functional status) EORTC IL353 measure (custom measure for this protocol) (fatigue, body image, financial toxicity). A higher score indicates greater fatigue, poorer body image and greater financial toxicity.
PRO: Difference over time in HRQoL (functional and aesthetic outcomes, fatigue, body image, financial toxicity) between Arm A and Arm B. | From allocation to 3-, 6-, 12-, 24- and 60 months median follow-up post-surgery.
  To determine the difference in breast-specific symptoms, cosmetic status, arm- and shoulder functional status measured by the BCTOS; and fatigue, body image, financial toxicity measured by the EORTC IL353between Arm A and Arm B.
PRO: Quality of Life Years (QALYs) between Arms A and Arm B. | At a median of 24 months follow up post-surgery.
  To determine the Quality of Life Years (QALYs) between Arms A and Arm B measured by the EQ-5D-5L. A high score indicates more problems.
PRO: Difference in QALYs over time between Arm A and Arm B. | From registration to allocation, 3-, 6-, 12-, 24- and 60 months median follow-up post-surgery..
  To determine the Quality of Life Years (QALYs) between Arms A and Arm B over time measured by the EQ-5D-5L. A high score indicates more problems.
PRO: Difference in Decision Regret between Arm A and Arm B. | At median of 24 months follow up post-surgery.
  To determine the difference in decision regret between Arm A and Arm B measured by Decision Regret Scale. A higher score indicates more regret.
PRO: Decision Regret in Arm A. | At median 24 months of follow-up post-surgery.
  To determine decision regret in Arm A measured by Decision Regret Scale. A higher score indicates more regret.
PRO: Overall mental health and depression over time between Arm A and Arm B. | From allocation to 3-, 6-, 12-, 24- and 60 months median follow-up post-surgery.
  To determine the overall mental health and differences over time in depression between Arm A and Arm B. Measured by the Patient Health Questionnaire-2. A higher score indicates and greater symptom burden.
PRO: Overall mental health and differences over time in anxiety in Arm A. | At 24 months median follow-up post-surgery.
  To determine the overall mental health and differences over time in anxiety in Arm A, measured by the Generalized Anxiety Disorder-2. A higher score indicates a higher symptom burden.
PRO: Overall mental health (depression) over time between Arm A and Arm B. | From allocation to 3-, 6-, 12-, 24- and 60 months median follow-up post-surgery.
  To determine the overall mental health and differences over time in depression between Arm A and Arm B. Measured by the Patient Health Questionnaire-2. A higher score indicates and greater symptom burden.
PRO: Overall mental health (anxiety) over time between Arm A and Arm B. | From allocation to 3-, 6-, 12-, 24- and 60 months median follow-up post-surgery.
  To determine the overall mental health and differences over time in anxiety between Arm A and Arm B. Measured by the Generalized Anxiety Disorder-2. A higher score indicates and greater symptom burden.

OTHER OUTCOMES:
ET: Oncologic outcomes in relation to intensity of endocrine therapy (ET) | Median of 5 and 10 years follow up
  To analyse oncological outcomes in relation to the intensity of endocrine therapy (ET) (no ET, less than 2 years ET, 2-5 years ET, more than 5 years ET).
Endocrine Therapy: Adherence to ET | Measured at a median of 6-, 24- and 60- months follow-up post-surgery.
  ET side effects as measured with the FACT-ES.
Radiology: Outcomes of MRI | At the time of the pre-operative MRI
  Outcomes of MRI in those patients who have MRI post-registration measured by BPR, occult lesion rate, biopsy approach, result of biopsy, malignant occult lesion rate.
Radiology: Occult lesion and malignant occult lesion detection rate | At the time of the pre-operative MRI
  To number of occult lesions and malignant occult lesions detected on pre-operative MRI per institution
Radiology: Frequency and nature of occult lesions from Contrast Enhanced Mammography (CEM) | At the time of the pre-operative MRI
  Measured by the frequency of occult lesions on CEM in patients undergoing CEM in addition to MRI and comparison of CEM and MRI findings.
Health Economics: The impact of the PROSPECTIVE model of care on costs and QALYs | 60-months post-surgery
  Health economic impact of including preoperative MRI and post-operative modification of adjuvant therapy in early breast cancer management in patients who have not had an MRI or CEM before PROSPECTIVE registration, as measured by QALYs (from the EQ-5D-5L).
Translational Research: Identify potential biomarkers of response and investigate tumour dynamics to identify patients in whom adjuvant therapy may be safely omitted. | At the time of diagnosis
  By sequencing and analysis of index tumours.
Translational Research: Identify potential biomarkers of response and investigate tumour dynamics to identify patients in whom adjuvant therapy may be safely omitted. | At the time of surgery for recurrence
  By sequencing and analysis of recurrent tumours.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Mann, MD, Study Chair — Melbourne Health; Steven David, MD, Study Chair — Peter MacCallum Cancer Centre - Moorrabin; Alastair Thompson, MD, Study Chair — Baylor College of Medicine
Locations (9):
- United States (2):
  - UCSF Breast Care Center, San Francisco, California
  - Baylor St Luke's Medical Centre, Houston, Texas
- Australia (7):
  - The Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - Mater Hospital, Sydney, North Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Cancer Centre (MMC Moorabbin), Clayton, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Anonymised Individual Patient Data (IPD) collected during the trial.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be made available for request after publication of the main/final study results; no end date.
Access Criteria: Researchers who submit a research proposal and BCT Data Request Application, which is assessed by BCT to have appropriate scientific value. Applications will be subject to approval by Breast Cancer Trials concept@bctrials.org.au (refer to BCT Data Sharing Guidelines).